CLINICAL TRIAL: NCT00995306
Title: A Double-Blind, Randomized, Controlled, Parallel-Group, Multicenter Study Evaluating the Safety and Efficacy of Civamide Cream 0.075% as a Treatment in Subjects With Osteoarthritis of the Knee
Brief Title: Evaluating the Safety and Efficacy Civamide in Osteoarthritis (OA) of the Knee(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Winston Laboratories (Industry)
Responsible Party: Scott B. Phillips, M.D., Study Director, Winston Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WL-1001-05-01; OA of the knee
Record Dates: First submitted 2008-02-25; First posted 2009-10-15 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis of the Knee
Keywords: Active comparator; Active civamide cream, 0.075%; Active civamide cream, 0.01%
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — zucapsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Civamide Cream 0.075%
  Interventions: Drug: Civamide (Zucapsaicin)
- 2 (Active Comparator): Civamide Cream 0.01%
  Interventions: Drug: Civamide (Zucapsaicin)

INTERVENTIONS:
Drug: Civamide (Zucapsaicin) — Civamide Cream 0.075%, TID for 12 weeks
  Civamide Cream 0.01%, TID for 12 weeks
  Other Names: Civamide; Zucapsaicin

SUMMARY:
To evaluate the safety and efficacy of Civamide Cream 0.075% as a treatment of the signs and symptoms associated with osteoarthritis of the knee.

DETAILED DESCRIPTION:
To ensure that both subjects and investigators remain blinded, the following design will be employed:

1. Subject Blinding: Randomization Subjects will be blinded to assignment to the placebo or active study drug: One half of the subjects will be randomized to Civamide Cream 0.075% to be applied on the Target Knee 3 times daily for 84 days (12 weeks). The other half will be randomized to Placebo Cream to be applied on the Target Knee 3 times daily for 84 days (12 weeks).

   As both Civamide Cream 0.075% and Placebo Cream can initially produce burning and stinging in some subjects, blinding to treatment assignment will be maintained. As the study progresses, the frequency of burning and stinging of both Civamide Cream 0.075% and Placebo Cream are expected to substantially decrease and be similar.
2. Investigator Blinding: Separate Raters To further maintain the blind, there will be two separate study staff raters: the Efficacy Rater Physician must be a physician-investigator who will evaluate efficacy parameters. The Safety Rater Physician must also be a physician-investigator who will evaluate safety parameters. A physician-investigator is defined as a physician who is listed as Principal Investigator or Sub-Investigator on Form FDA 1572. Each may assign a designee (another appropriately trained study staff member) to perform study procedures (as defined in Section 8.0 or Appendix E, for the Study Staff Responsibility Chart).

Study Periods:

See Study Flow Chart and Schedule of Observations.

Screening Period (Day -3):

The following procedures will be conducted: Obtain informed consent; assess eligibility according to selection criteria; collect demographic data, medical history, osteoarthritis history and diagnosis, and prior and current medications information. Perform physical examination and obtain vital signs and laboratory tests (chemistry, hematology & urinalysis). Female subjects of child-bearing potential will be given a urine pregnancy test. The subject will complete the Screening Pain Scale for both knees. Either Rater Physician will determine the subject's Functional Capacity Classification. If the subject is eligible, (i.e., Screening Pain Subscale score of ≥ 9 in one knee, subject does not have regular, significant pain due to OA or other conditions in the other knee, and has a Functional Capacity Classification score of I-III) the Efficacy Rater Physician or Safety Rater Physician will identify the knee joint with the most severe symptoms of OA as the "Target Knee". The subject must have an x-ray or radiographic report available within the last 3 years in order to meet the Selection Criteria. If the subject has no prior x-ray or radiographic report an x-ray of the Target Knee will be obtained.

Baseline/Randomization Period (Day 1) Either Rater Physician will review laboratory test and x-ray results of the Target Knee prior to randomization and confirm subject's continued eligibility including compliance with stability of the oral NSAIDs/COX-2 medications prior to randomization.

Subjects will complete another Screening Pain Scale to confirm that the Target Knee score is > 9. If eligible, the subject will be randomized into the Double-Blind Treatment Period.

If the Screening Pain Scale score is less than 9, the subject may return within 14 days of the first clinic visit (Visit 1/Day -3) to repeat it. If eligible at that time, the scheduled Baseline procedures will be performed and completed.

Eligible subjects will complete the WOMAC OA Index, the Subject's Global Evaluation, and the SF-36® Health Survey.

Subjects will apply their first dose of study drug in the clinic. They will be sent home with diaries to complete everyday, and with study drug that will be applied only on the Target Knee three times daily.

Treatment Period (Days 1-84):

The subject will complete the WOMAC OA Index and Subject's Global Evaluation at clinic visits on Days 1, 21, 42, 63 and 84 (not Day 3). Concurrent medications, adverse events, and study drug compliance will be reviewed and recorded by the Safety Rater Physician or designee throughout the Treatment Period at clinic visits on Days 3, 21, 42, 63 and 84 (End-of-Study/Final Visit).

Also on Day 84 (End-of-Study/Final Visit), the subject will complete the SF-36® Health Survey, the Efficacy Rater Physician will determine the Functional Capacity Classification, the Safety Rater Physician or designee will complete a final set of vital signs and collect laboratory samples. The Safety Rater Physician will perform a complete physical examination on each subject and will review laboratory results when available.

Safety Rater Physician or designee will contact the subject by phone on Days 15, 36, 57 and 78 to assess subject compliance with study drug application, maintenance of concurrent medications, including stable dose of NSAIDS or COX-2 inhibitors, review adverse events experienced, determine if subject has enough study drug to last until the next visit, and remind the subject of the next scheduled clinic visit.

On Day 84 (End-of-Study/Final Visit) the subject will be discharged after all procedures have been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an IRB-approved informed consent prior to entry into the Screening Period (Day -3).
2. Subject has OA pain of the Target Knee with a WOMAC Pain Subscale baseline value of > 9 at the Baseline/Randomization Period (Maximum score is 20 for 5 questions with 0 = none; 4 = extreme.
3. Subject must have a Functional Capacity Classification of I-III.
4. Subject has taken a stable dose of NSAIDs or COX-2 inhibitor agents for OA pain for at least 22 of the previous 28 days and for each of the 2 days prior to the Screening Period (Day -3) and for at least each of the 2 days prior to the Baseline/Randomization Period (Day 1). Subject must also, agree and be expected to remain on this stable daily dose throughout the study.
5. Subject is between 40-75 years of age.
6. Diagnosis of OA is present for at least 6 months according to the ACR criteria for OA of the knee.
7. Radiographic evidence of OA of the Target Knee (within the last 3 years) with a Kellgren-Lawrence scale of 2 or 3.
8. Subject is generally in good health.
9. Subject is expected to be compliant with study procedures.
10. Females of child-bearing potential must have a negative urine pregnancy test at Screening.
11. Female subjects of child-bearing potential agree to use an approved form of contraception and must be on the same contraceptive method and dosage schedule during the entire study.

Exclusion Criteria:

1. Presence of tendonitis, bursitis, partial or complete joint replacement of Target Knee.
2. Presence of active skin disease, erythema, infection, wound or irritation near the treatment area of the Target Knee.
3. Subject has history of frequent headache or other painful conditions (other than OA) that is expected to require any use of systemic opiates or derivatives, or more than twice a week additional administration of different oral NSAIDs or COX-2 inhibitors (see Section 6.1, Table 2).
4. Subject experiences regular significant pain due to osteoarthritis or other conditions in the non-target knee or other joints while on stable doses of their current analgesic therapy.
5. Subject has an anticipated need for any surgical or other invasive procedure that will be performed on the Target Knee or other part of the body during the course of the study.
6. OA secondary to local joint disorders (e.g., mechanical disorder, internal derangement of the knee), systemic metabolic disease, endocrine disorders, bony dysplasia, calcium crystal deposition disease, neuropathic arthropathy, frostbite, congenital abnormalities.
7. Subject has history and/or diagnosis of rheumatoid arthritis, fibromyalgia, connective tissue disease, psoriatic arthritis, erosive inflammatory OA, diffuse idiopathic skeletal hyperostosis, severe neurologic or vascular disease.
8. Subject has active (redness, swelling, fever, etc.) gout/pseudogout within 6 months prior to screening.
9. Subject has Type I or Type II diabetes with peripheral neuropathies.
10. Subject is extremely obese with BMI ≥ 39.
11. Subject has had trauma to or surgery on the Target Knee within 1 year of Screening/Baseline.
12. Subject has an underlying clinical condition, including previous malignancies that in the Investigator's judgment, is unstable.
13. Subject has known allergy or hypersensitivity to capsicum, civamide, or capsaicin-containing products or any constituent of the cream formulation.
14. Subject has a history of substance abuse within the past 12 months.
15. Subject has participated in previous clinical study with Civamide Cream.
16. Use of restricted medications (See Medication/Treatment Table, Section 5.1.2).

Ages: 40 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2003-06; Primary Completion 2004-04 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain
WOMAC Physical Function
Subject's Global Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Phillips, M.D., Study Director — Winston Laboratories